CLINICAL TRIAL: NCT02995889
Title: FLT-PET for Early Detection of Relapse in Patients With Irradiated Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Tine Nøhr Christensen, MD, research fellow, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 308_14
Record Dates: First submitted 2016-12-09; First posted 2016-12-19 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-05

CONDITIONS: Lung Cancer, Nonsmall Cell; Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

ARMS (1):
- FLT-PET (Experimental)
  Interventions: Device: FLT-PET

INTERVENTIONS:
Device: FLT-PET

SUMMARY:
This study investigates the feasibility of FLT-PET to improve the diagnosis of relapse in patients with irradiated lung cancer in comparison with FDG-PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* history with lung cancer, small cell or non-small cell
* radiotherapy of lung cancer ended within the last 24 months
* radiotherapy might be normofractionated or stereotactic
* current suspicion of relapse
* written and oral consent

Exclusion Criteria:

* communication difficulties
* pregnancy or lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-11; Primary Completion 2019-02-07 (Actual); Study Completion 2020-02-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with local and/or regional relapse | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Kjær, MD phD MDSci, Study Chair — Dept of Clinical Physiology, Nuclear medicine and PET, Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Dept. of Clinical Physiology, Nuclear Medicine and PET, Rigshospitalet, Copenhagen
  - Dept. Respiratory Medicine, Bispebjerg University Hospital, Copenhagen

REFERENCES:
- [Result] Christensen TN, Langer SW, Persson G, Larsen KR, Loft A, Amtoft AG, Berthelsen AK, Johannesen HH, Keller SH, Kjaer A, Fischer BM. 18F-FLT PET/CT Adds Value to 18F-FDG PET/CT for Diagnosing Relapse After Definitive Radiotherapy in Patients with Lung Cancer: Results of a Prospective Clinical Trial. J Nucl Med. 2021 May 10;62(5):628-635. doi: 10.2967/jnumed.120.247742. Epub 2020 Oct 9. PMID 33037090
- [Result] Christensen TN, Langer SW, Persson G, Larsen KR, Amtoft AG, Keller SH, Kjaer A, Fischer BM. Impact of [18F]FDG-PET and [18F]FLT-PET-Parameters in Patients with Suspected Relapse of Irradiated Lung Cancer. Diagnostics (Basel). 2021 Feb 11;11(2):279. doi: 10.3390/diagnostics11020279. PMID 33670242